CLINICAL TRIAL: NCT03954626
Title: A Single-Arm, Open-Label, Multicenter, Phase IIIb Study to Collect Safety and Electrocardiogram Data on Brolucizumab 6 mg Intravitreal Treatment in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Study to Collect Safety and ECG Data on Brolucizumab 6 mg Intravitreal Treatment in Patients With Wet AMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTH258A2309
Record Dates: First submitted 2019-05-08; First posted 2019-05-17 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-08

CONDITIONS: Age-Related Macular Degeneration; Macular Degeneration; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases
Keywords: AMD, nAMD, wet AMD, RTH258, brolucizumab, ECG, open-label
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases | interventions — brolucizumab

STUDY DESIGN:
Intervention Model Description: Single arm, multicenter
Masking Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RTH258 (Experimental): Intravitreal injection
  Interventions: Biological: brolucuzumab 6 mg IVT

INTERVENTIONS:
Biological: brolucuzumab 6 mg IVT — Single intravitreal injection (IVT) of brolucizumab 6 mg
  Other Names: RTH258

SUMMARY:
The purpose of this study was to collect ECG data after a single IVT injection of brolucizumab 6 mg in patients with neovascular age-related macular degeneration (nAMD).

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter study that collected ECG data after a single IVT injection of brolucizumab 6 mg in patients with nAMD. Triplicate 12-lead ECG recording was performed at screening to determine eligibility. A second triplicate 12-lead ECG recording was collected approximately 2h prior to the brolucizumab IVT injection on Day 1. Holter ECG recording started approximately 1 h prior to the brolucizumab IVT injection and ended approximately 48h after the IVT injection. A third triplicate 12-lead ECG recording was performed after the conclusion of Holter monitoring on Day 3.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent MUST be obtained prior to participation in the study
* Study eye is diagnosed with nAMD and deemed to be eligible for intravitreal injection at the discretion of the Investigator

Exclusion Criteria:

* Concomitant conditions or ocular disorders in the study eye at screening which may cause safety concerns on the judgement of the investigator
* Any active intraocular or periocular or systemic infection or active intraocular inflammation at Baseline
* Treatment with any ocular intravitreal injection in the study eye within the past 7 half lives prior to Baseline
* Intraocular surgery, prior long-acting therapeutic agent, or ocular drug release device implantation (approved or investigational) in the study eye any time during the past 3 months prior to Baseline
* Diagnosis of ECG abnormalities including:
* Clinically significant cardiac arrhythmias, e.g., atrial fibrillation, sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker
* Familial long QT syndrome or known family history of Torsades de Pointes
* Resting heart rate < 50 or > 90 bpm at screening
* Resting QTcF ≥ 450 ms (male) or ≥ 460 ms (female) at screening
* Use of concomitant medications that are classified as known risk, conditional risk or possible risk to prolong QT/QTc interval within 7 half-lives prior to Baseline
* History of stroke (including transient ischemic attack, reversible ischemic neurological deficit, prolonged reversible ischemic neurological deficit) or myocardial infarction (ST or non-ST elevation myocardial infarction) at any time prior to baseline
* Chronic kidney disease as determined as a CrCL at screening of < 60 ml/min/1.73 m2 as determined by the MDRD formula
* Uncontrolled high blood pressure defined as a systolic value ≥ 140 mmHg or diastolic value ≥ 90 mmHg at screening or baseline
* Systemic anti-VEGF therapy during the 6-month period prior to baseline
* Electrolyte disturbances determined as out of normal range sodium, potassium or calcium serum concentrations at screening
* Concomitant intake of long-acting muscarinic antagonist (LAMA)/ long-acting beta adrenergic (LABA) combination therapy
* History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar classes as assessed by the investigator
* Use of systemic or ocular (including intravitreal) investigational drugs within 7 half-lives of baseline, (or within 30 days/until the expected pharmacodynamic effect has returned to baseline), whichever is longer or longer if required by local regulations (observational clinical studies solely involving over-the-counter vitamins, supplements, or diets are not exclusionary)
* Pregnant or nursing (lactating) women

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Zakaria, MD, Study Director — Novartis Institutes for BioMedical Research
Locations (3):
- United States (2):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Abilene, Texas
- Novartis Investigative Site, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Zakaria N, Guerard N, Emanuelli A, Dugel P, Watts J, Liew M, Gekkieva M, Hinder M. Evaluation of cardiac parameters and other safety outcomes of brolucizumab treatment in patients with neovascular age-related macular degeneration. Pharmacol Res Perspect. 2022 Apr;10(2):e00897. doi: 10.1002/prp2.897. PMID 35301822
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled patients from 3 centers from the United States.14 patients were enrolled and analyzed in the study.
Period: Overall Study
Arm/Group | RTH258
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Fourteen patients were enrolled at 3 sites in the US, all of which completed the study
Arm/Group | RTH258
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.7 (6.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Clinically Relevant Treatment Emergent ECG Changes After Intravitreal Injection of Brolucizumab 6 mg in Patients With nAMD
Description: Incidence between 20 and 24 h post-injection of clinically relevant treatment emergent changes in heart rate (HR), pulse rate (PR), QRS, and QTc (heart rate corrected QT using Fridericia's formula, QTcF) interval (ms). This is a composite endpoint capturing all 4 parameters and 3 time-points in one Outcome Measure.
Time Frame: Baseline, Hour 20, Hour 22, Hour 24
Population: The safety analysis, which included all patients who received one intravitreal injection of brolucizumab 6 mg.
Measure: Number; unit: Number of events
Arm/Group | RTH258
Number analyzed (Participants) | 14
Number of events | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from date of written informed consent until the end of study visit (Day 8)
Arm/Group | RTH258
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RTH258 (N=14)
Intraocular pressure increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT03954626/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT03954626/SAP_001.pdf